CLINICAL TRIAL: NCT03204643
Title: An Evaluation of ED to Admission Conversion Among Patients With a Telepsychiatric Consult Who Are Followed by a Behavioral Health - Virtual Patient Navigation Team
Brief Title: Evaluation of Behavioral Health-Virtual Patient Navigation Team (BH-VPN)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 00021808
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Results first posted 2019-10-02 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2020-01

CONDITIONS: Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BH-VPN (Experimental): A bundle of usual care components applied consistently and completely, plus access to mental health trained patient navigators and navigation services.
  Interventions: Behavioral: BH-VPN
- Usual Care (No Intervention): The standard intervention (Control - Usual Care) is given in this population. May contain some of the BH-VPN components.

INTERVENTIONS:
Behavioral: BH-VPN — A bundle of usual care components, applied consistently and completely, along with access to behavioral health specific patient navigators and navigation services.
  Arms: BH-VPN

SUMMARY:
Patients who present to one of the participating EDs with a telepsychiatric consult performed will be treated and followed per the behavioral health virtual patient navigation pathway (BH-VPN) or usual care. The BH-VPN is inclusive of several components which will all be consistently applied to patients randomized to the intervention, as well as having access to behavioral health trained patient navigators. These key components are often deployed inconsistently as a part of usual care, but per the intervention, will be completed in totality for subjects who are assigned to and participate in the BH-VPN plan.

This study includes a qualitative sub-study to measure perceptions of the impact of the BH-VPN on readmission rates and patient outcomes, experiences with the services provided by the BH-VPN, and provider and clinician ideas for how to improve the services provided by the BH-VPN.

ELIGIBILITY:
Inclusion Criteria:

* Present at a participating ED
* Completed telepsychiatric consult as captured in the EMR
* Completed telepsychiatric consult Monday - Friday during Navigator's potential hours of operation.

Exclusion Criteria:

* None per the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 637 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2018-02-14 (Actual); Study Completion 2018-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Sparks, MD, Principal Investigator — Wake Forest University Health Sciences; Jason Roberge, PhD, Study Director — Wake Forest University Health Sciences
Locations (6):
- United States (6):
  - Carolinas Medical Center Mercy, Charlotte, North Carolina
  - Carolinas Healthcare System - Pineville, Charlotte, North Carolina
  - Carolinas Healthcare System University, Charlotte, North Carolina
  - Carolinas Healthcare System Steele Creek, Charlotte, North Carolina
  - Carolinas Healthcare System Huntersville, Huntersville, North Carolina
  - Carolinas Healthcare System - Union, Monroe, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roberge J, McWilliams A, Zhao J, Anderson WE, Hetherington T, Zazzaro C, Hardin E, Barrett A, Castro M, Balfour ME, Rachal J, Krull C, Sparks W. Effect of a Virtual Patient Navigation Program on Behavioral Health Admissions in the Emergency Department: A Randomized Clinical Trial. JAMA Netw Open. 2020 Jan 3;3(1):e1919954. doi: 10.1001/jamanetworkopen.2019.19954. PMID 31995214

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BH-VPN | Usual Care
Started (All those randomized to the intervention were included in the analysis) | 323 | 314
Completed | 323 | 314
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BH-VPN | Usual Care | Total
Number analyzed (Participants) | 323 | 314 | 637
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (16.8) | 39.8 (16.3) | 39.7 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 139 | 279
  Male | 183 | 175 | 358
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 105 | 90 | 195
  White | 170 | 182 | 352
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 39 | 37 | 76
Region of Enrollment [Number; unit: participants]
  United States | 323 | 314 | 637

OUTCOME MEASURES:

1. Primary Outcome: Emergency Department to Inpatient Conversion Rate
Description: admission from the Emergency Department with behavioral health consult completed, to an inpatient or observation setting.
Time Frame: 5 days
Population: The number of patients that were admitted
Measure: Number; unit: participants
Arm/Group | BH-VPN | Usual Care
Number analyzed (Participants) | 323 | 314
participants | 178 | 198
Statistical Analysis 1: Comparison: BH-VPN vs Usual Care; Test type: Superiority; p = 0.06, Regression, Logistic; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.54 to 1.02]

2. Secondary Outcome: Quality, Comfort, and Care (QCC) Defined Readmission Rate
Description: readmission within 30 days to the same facility
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | BH-VPN | Usual Care
Number analyzed (Participants) | 323 | 314
Participants | 7 | 2
Statistical Analysis 1: Comparison: BH-VPN vs Usual Care; Test type: Superiority; p = 0.76, Mixed Models Analysis; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.70 to 1.64]

3. Secondary Outcome: Patient-centric (Protocol Defined) Readmission Rate
Description: readmission within 30 days to any facility which Carolinas Healthcare System have access to the data
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | BH-VPN | Usual Care
Number analyzed (Participants) | 323 | 314
Participants | 28 | 23
Statistical Analysis 1: Comparison: BH-VPN vs Usual Care; Test type: Superiority; p = 0.62, Mixed Models Analysis; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.65 to 2.08]

4. Secondary Outcome: Utilization of Healthcare Services Post-discharge From Emergency Department
Description: Number of Emergency Department, inpatient, observation encounters
Time Frame: 45 days
Measure: Count of Participants; unit: Participants
Arm/Group | BH-VPN | Usual Care
Number analyzed (Participants) | 323 | 314
Participants | 112 | 89
Statistical Analysis 1: Comparison: BH-VPN vs Usual Care; Test type: Superiority; p = 0.08, Mixed Models Analysis; Odds Ratio (OR) = 1.35, 0.96% CI 2-sided [0.96 to 1.90]

ADVERSE EVENTS:
Time Frame: We followed each patient for 45 days after the ED discharge and then followed the patient for an additional 60 days for utilization outcomes.
Arm/Group | BH-VPN | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/323 | 4/314
Serious Adverse Events (participants affected / at risk) | 0/323 | 0/314
Other Adverse Events (participants affected / at risk) | 0/323 | 0/314

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/43/NCT03204643/Prot_SAP_000.pdf